CLINICAL TRIAL: NCT04484116
Title: USEFULNESS OF IOPTH AS A PREDICTOR FOR SUCCESSFUL PARATHYROIDECTOMY IN SECONDARY HYPERPARATHYROIDISM: A COHORT STUDY
Brief Title: IOPTH Usefulness for Predicting Successful Surgery in Secondary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Hospital General Ajusco Medio (Other)
Responsible Party: Principal Investigator, Karla Verónica Chavez-Tostado, MD, Hospital General Ajusco Medio
Other Study IDs: Not assigned
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary hyperparathyroidism; Parathyroidectomy; Intraoperative paratohormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Succesful surgery: PTH 24 hours after surgery <150pg/mL
  Interventions: Diagnostic Test: Intraoperative Paratohormone
- Unsuccessful surgery: PTH 24 hours after surgery >150pg/mL
  Interventions: Diagnostic Test: Intraoperative Paratohormone

INTERVENTIONS:
Diagnostic Test: Intraoperative Paratohormone — Three IOPTH determinations were withdrawn: at anesthetic induction (PTH0), 15 minutes (PTH15), and 30 minutes (PTH30) after completion gland resection. Another sample was taken 24 hours after the procedure (PTH24), values <150pg/mL defined a successful surgery and patients were assigned to the successful or unsuccessful group. IOPTH drop was analyzed to predict successful surgery with drops of 70% and 90% at 15 and 30 minutes.

SUMMARY:
Secondary hyperparathyroidism (SHPT) is a multisystemic syndrome that affects calcium and bone homeostasis in patients with chronic kidney disease (CKD). Despite medical treatment, 1-2% of patients require parathyroidectomy anually. The use of an intraoperative paratohormone protocol (IOPTH) to predict cure still in debate, due to the lack of standardized protocols, the use of different assays and uneven PTH clearance. The aim of this study was to determine the diagnostic accuracy of an IOPTH in patients with SHPT for predicting successful surgery after parathyroidectomy.

DETAILED DESCRIPTION:
A prospective observational study (cohort) was performed in patients who were submitted to parathyroidectomy by an endocrine surgeon for SHPT. All were submitted to a bilateral neck exploration with a subtotal parathyroidectomy. Three IOPTH determinations were withdrawn: at anesthetic induction (PTH0), 15 minutes (PTH15), and 30 minutes (PTH30) after completion gland resection. Another sample was taken 24 hours after the procedure (PTH24), values <150pg/mL defined a successful surgery and patients were assigned to the successful or unsuccessful group. IOPTH drop was analyzed to predict successful surgery with drops of 70% and 90% at 15 and 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* PTH >800pg/mL and SHPT symptoms, or
* Asymptomatic patients with PTH >1000pg/mL who were resistant to treatment
* compliance with the signature of the informed consent

Exclusion Criteria:

* patients who respond adequately to medical treatment
* incomplete IOPTH protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease and secondary hyperparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Successful surgery | 24 hours
  Biochemical response to subtotal prathyroidectomy

SECONDARY OUTCOMES:
PTH drop | 15 minutes and 30 minutes after resection
  Drop from baseline, aiming a drop >70%

CONTACTS AND LOCATIONS:
Overall Officials: Karla V Chavez-Tostado, MD, Principal Investigator — SEDESA
Locations (1):
- Hospital General Ajusco Medio, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pitt SC, Sippel RS, Chen H. Secondary and tertiary hyperparathyroidism, state of the art surgical management. Surg Clin North Am. 2009 Oct;89(5):1227-39. doi: 10.1016/j.suc.2009.06.011. PMID 19836494
- [Result] IV. NKF-K/DOQI Clinical Practice Guidelines for Anemia of Chronic Kidney Disease: update 2000. Am J Kidney Dis. 2001 Jan;37(1 Suppl 1):S182-238. doi: 10.1016/s0272-6386(01)70008-x. No abstract available. PMID 11229970
- [Result] Young EW, Albert JM, Satayathum S, Goodkin DA, Pisoni RL, Akiba T, Akizawa T, Kurokawa K, Bommer J, Piera L, Port FK. Predictors and consequences of altered mineral metabolism: the Dialysis Outcomes and Practice Patterns Study. Kidney Int. 2005 Mar;67(3):1179-87. doi: 10.1111/j.1523-1755.2005.00185.x. PMID 15698460
- [Result] Lorenz K, Bartsch DK, Sancho JJ, Guigard S, Triponez F. Surgical management of secondary hyperparathyroidism in chronic kidney disease--a consensus report of the European Society of Endocrine Surgeons. Langenbecks Arch Surg. 2015 Dec;400(8):907-27. doi: 10.1007/s00423-015-1344-5. Epub 2015 Oct 2. PMID 26429790
- [Result] Carneiro DM, Solorzano CC, Nader MC, Ramirez M, Irvin GL 3rd. Comparison of intraoperative iPTH assay (QPTH) criteria in guiding parathyroidectomy: which criterion is the most accurate? Surgery. 2003 Dec;134(6):973-9; discussion 979-81. doi: 10.1016/j.surg.2003.06.001. PMID 14668730
- [Result] Hruska KA, Korkor A, Martin K, Slatopolsky E. Peripheral metabolism of intact parathyroid hormone. Role of liver and kidney and the effect of chronic renal failure. J Clin Invest. 1981 Mar;67(3):885-92. doi: 10.1172/jci110106. PMID 7204561
- [Result] Hiramitsu T, Tominaga Y, Okada M, Yamamoto T, Kobayashi T. A Retrospective Study of the Impact of Intraoperative Intact Parathyroid Hormone Monitoring During Total Parathyroidectomy for Secondary Hyperparathyroidism: STARD Study. Medicine (Baltimore). 2015 Jul;94(29):e1213. doi: 10.1097/MD.0000000000001213. PMID 26200645
- [Result] Seehofer D, Rayes N, Klupp J, Steinmuller T, Ulrich F, Muller C, Schindler R, Frei U, Neuhaus P. Predictive value of intact parathyroid hormone measurement during surgery for renal hyperparathyroidism. Langenbecks Arch Surg. 2005 Jun;390(3):222-9. doi: 10.1007/s00423-005-0541-z. Epub 2005 Feb 22. PMID 15726399
- [Result] Vulpio C, Bossola M, Di Stasio E, Pepe G, Nure E, Magalini S, Agnes S. Intra-operative parathyroid hormone monitoring through central laboratory is accurate in renal secondary hyperparathyroidism. Clin Biochem. 2016 May;49(7-8):538-43. doi: 10.1016/j.clinbiochem.2016.01.012. Epub 2016 Jan 20. PMID 26800781
- [Result] Lokey J, Pattou F, Mondragon-Sanchez A, Minuto M, Mullineris B, Wambergue F, Foissac-Geroux P, Noel C, de Sagazan HL, VanHille P, Proye CA. Intraoperative decay profile of intact (1-84) parathyroid hormone in surgery for renal hyperparathyroidism--a consecutive series of 80 patients. Surgery. 2000 Dec;128(6):1029-34. doi: 10.1067/msy.2000.110431. PMID 11114639
- [Result] Barczynski M, Cichon S, Konturek A, Cichon W. A randomised study on a new cost-effective algorithm of quick intraoperative intact parathyroid hormone assay in secondary hyperparathyroidism. Langenbecks Arch Surg. 2005 Apr;390(2):121-7. doi: 10.1007/s00423-004-0535-2. Epub 2005 Feb 15. PMID 15711996